CLINICAL TRIAL: NCT01460927
Title: Clinical Study to Evaluate the Performance of TriActive+ RF for the Non-invasive Treatment of Wrinkles & Rhytides
Brief Title: TriActive+ Radiofrequency (RF) for Non-invasive Treatment of Wrinkles & Rhytides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deka Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TriActive+RF-DEKA-092011
Record Dates: First submitted 2011-10-24; First posted 2011-10-27 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Wrinkles; Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TriActive+ RF (Other): Healthy male or female subjects 30-60 years of age, having at least two facial sub-areas (left peri-orbital, right peri-orbital or peri-oral) with visible lines/wrinkles and elastosis, which correlate to a score of 2-6 on the Fitzpatrick Classification of Wrinkling and Degree of Elastosis.
  Interventions: Device: TriActive+ RF

INTERVENTIONS:
Device: TriActive+ RF — Radio frequency handpiece uses a multi-polar technology with a particular electrical frequency of 1MHz. The handpiece has a special "skin contact identification" system which delivers energy only when electrodes are adherent to the skin surface in order to avoid the prickling sensation when the treatment starts.

SUMMARY:
The study objective is to evaluate the safety and efficacy of a radiofrequency (RF) source, the TriActive+ RF handpiece, for treatment of wrinkles and rhytides after multiple treatments. The primary endpoint is observation of changes to the surface by visual and photographic analysis. Secondary endpoints: measurement of patient satisfaction and comfort of the treatment and the measurement of adverse events.

DETAILED DESCRIPTION:
Collagen varies genetically and structurally. Collagen breakdown increases with chronological age and photoaging. While fibroblasts normally replace damaged collagen fibers with new ones, the ability of fibroblasts to replace collagen is compromised by natural aging and environmental stress. Although collagen fibers form a loose interlacing network that is deformable, increased collagen breakdown leads to thinning and loss of the elastic fiber network in the dermis. This breakdown results in the formation of wrinkles, especially in areas of the skin exposed to the sun, which are most prone to wrinkles and imperfections. Nonablative dermal remodeling has gained tremendous popularity among patients and practitioners, offering a low incidence of adverse effects and modest improvement in the various signs of cutaneous photoaging, including rhytides, dyschromias and telangiectasias. Controlled thermal skin injury has been shown to effect a conformational change in the structure and length of collagen and may also induce fibroblast response for long-term collagen remodeling. Interest in utilizing radiofrequency energy to enhance deep tissue tightening and thus improve skin laxity has grown, as radiofrequency energy has been shown in multiple studies to tighten tissue, producing a noticeable skin lifting.

This study is intended to evaluate the clinical performance of a radiofrequency (RF) source as engendered in the TriActive+ RF for the non-invasive treatment of wrinkles and rhytides.

Eligible subjects who have signed an ICF will receive up to 8 treatments on at least two facial sub areas (left peri-orbital, right peri-orbital and peri-oral). Up to 25 subjects will be enrolled in the study. Treatments will start at a low power and then gradually increase, based on tolerability and tissue reaction. The goal is to progressively reach and maintain an epidermal temperature end-point. The site will use an IR thermometer to ensure the rise in temperature does not exceed 42° C.

Treatments will be once a week with follow-up visits at one week, one month, and three months following the final treatment. Clinical assessments by the investigator and digital photographs will be taken prior to the baseline treatment, immediately prior to the 4th and 8th treatment, and at the 1 month and 3 month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent agreement signed by the subject.
* Healthy male or female subjects 30-60 years of age.
* Having at least two facial sub-areas (left peri-orbital, right peri-orbital or peri-oral) with visible lines/wrinkles and elastosis, which correlate to a score of 2-6 on the Fitzpatrick Classification of Wrinkling and Degree of Elastosis.
* Willingness to follow the treatment and follow-up schedule and the post-treatment care.
* For female candidates - post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).

Exclusion Criteria:

* Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breastfeeding.
* Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
* Having a permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.
* Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session.
* Use of retinoids, antioxidants or skin nourishing supplements within 1 month of treatment or during the study.
* Having received a facial within 1 month of treatment or during the study.
* Having received a facial dermabrasion or chemical peel treatment within 2 months of treatment or during the study.
* Having received treatment with light, RF or other devices in the treated area within 6 months of treatment or during the study.
* Having received Botox in the treated area within 6 months of treatment or during the study.
* Having received collagen/Hyaluronic Acid (HA) in the treated area within a year of treatment or during the study.
* Having undergone a resurfacing procedure, face lift or eyelid surgery within a year of treatment or during the study.
* Having undergone any other surgery in the treated area within 6 months of treatment (or more if skin has not healed completely) or during the study.
* Having ever received fat injections or other methods of augmentation with injected or implanted material in the treated area or planning to during the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Gabriel, MD, Principal Investigator — Southwest Medical Group Plastic Surgery
Locations (1):
- Southwest Medical Group Plastic Surgery, Vancouver, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TriActive+RF: Subjects will receive up to 8 treatments on at least two facial sub areas (e.g., left peri-orbital, right peri-orbital and/or peri-oral). Treatments will be administered once a week (±2days) with evaluation follow-up visits at one (1) week (±2days), one (1) month (±4days), and three (3) months (±4days) following the final treatment. The treatments start at a low power (3W for the small tip, 10W for the medium and large tips) and then gradually increase the setting up to the highest powers available within the tips, checking the subject's tolerability and reaction of the tissue.
  The power is adjusted to suit the subject's sensitivity and the "depth" of tissue to be treated (deeper tissue requires the larger tip). The goal is to progressively and smoothly reach an epidermal temperature end-point of 43°C. The treatment end-point correlates directly with the measurement of the skin temperature.
  The temperature of 43°C should be maintained at the end point for several minutes (3-5min).
Period: Overall Study
Arm/Group | TriActive+RF
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TriActive+ RF
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Fitzpatrick Classification of Wrinkling and Degree of Elastosis.
Description: At each of the specified time points, photographs of the treated areas will be taken. The photography angles will include a global frontal photo and the right and left sides of the face at 45° and/or 90°. In addition, close up photos will be taken of specific facial zones, e.g., the peri orbital wrinkles.
  Observing changes to the surface by visual and photographic analysis based on the score of 2-6 on the Fitzpatrick Classification of Wrinkling and Degree of Elastosis. (Lasers Surg Med 2003;33(4):232 42)
  Score Wrinkling & Degree of Elastosis 1-3 Fine wrinkles (rhytides) and Mild Elastosis (fine textural changes with subtly accentuated skin lines) 4-6 Fine to moderate depth wrinkles, moderate number of lines and Moderate Elastosis (distinct papular elastosis [individual papules with yellow translucency under direct lighting] and dyschromia)
Time Frame: Baseline, Pre Treatment 4, Pre Treatment 8, 1 Month FU, 3 Month FU
Population: Per protocol
Measure: Mean (Full Range); unit: Fitzpatrick Classification Scale
Groups:
- Baseline: Baseline (before Treatments)
- Pre Treatment 4: After 3 treatments
- Pre Treatment 8: After 7 treatments
- 1 Month FU: 1 Month after the 8th treatment
- 3 Month FU: 3 Months after the 8th treatment
Arm/Group | Baseline | Pre Treatment 4 | Pre Treatment 8 | 1 Month FU | 3 Month FU
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Fitzpatrick Classification Scale | 5.6 (1) [1 to 6] | 5.56 (2) [1 to 6] | 5.36 [1 to 6] | 5.32 [1 to 6] | 4.88 [1 to 6]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- TriActive+RF: Subjects will receive up to 8 treatments with the TriActive+ RF on at least two facial sub areas (e.g., left peri-orbital, right peri-orbital and/or peri-oral). Treatments will be administered once a week (±2 days).
Arm/Group | TriActive+RF
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TriActive+RF (N=25)
Irritation, itching, erythema, edema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall have the right to publish the results of the Trial provided Sponsor has given it prior written approval. Sponsor reserves the right to remove all Confidential Information from any communications, or if Sponsor deems that such removal does not sufficiently protect its intellectual property rights, to require that Investigator refrain from making such communications.